CLINICAL TRIAL: NCT03478826
Title: Creation of a Biospecimen Repository From Patients With Interstitial Lung Diseases (ILD)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eva M. Carmona Porquera, Assistant Professor of Medicine, College of Medicine, Mayo Clinic
Other Study IDs: 17-008088
Record Dates: First submitted 2018-03-23; First posted 2018-03-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Interstitial Lung Disease
Keywords: ILD
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — To develop a repository of blood samples from patients with ILD to support future studies into the development of such biomarkers. Patients with pneumonia and healthy patients will also be recruited as a control group. The repository would be maintained in Dr. Carmona's laboratory in the Thoracic Diseases Research Unit in the Stabile building where all biospecimens will be stored.
  These samples will be stored in freezers in Dr. Carmona's laboratory space in the Thoracic Diseases Research Unit in the Stabile building for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ILD: 250 patients (male and females >18 years of age) with the diagnosis of fibrotic DILD (IPF (n=100), fibrotic NSIP (n=50), chronic hypersensitivity pneumonia (n=20), sarcoidosis(n=50), progressive rheumatoid lung disease (n=10) and scleroderma lung disease (n=20), 10 patients with other fibrosing disease (fibrosing mediastinitis), and 50 patients with lymphangioleiomyomatosis.
  Interventions: Other: ILD
- Healthy: 100 healthy participants as a control group.
  Interventions: Other: Healthy
- Pneumonia: 25 patients with pneumonia as a control group.
  Interventions: Other: Pneumonia

INTERVENTIONS:
Other: ILD — 100 cc of blood collected from a total of 250 ILD patients. This includes IPF (n=100), fibrotic NSIP (n=50), chronic hypersensitivity pneumonia (n=20), sarcoidosis(n=50), progressive rheumatoid lung disease (n=10) and scleroderma lung disease (n=20)), 10 patients with other fibrosing disease (fibrosing mediastinitis), and 50 patients with lymphangioleiomyomatosis
  Groups: ILD
Other: Healthy — 100 cc of blood collected from a total of 25 healthy volunteers in order to compare with the ILD participants.
  Groups: Healthy
Other: Pneumonia — 100 cc of blood collected from a total of 100 participants with a diagnosis of pneumonia in order to compare with the ILD participants.
  Groups: Pneumonia

SUMMARY:
To develop a repository of blood samples from patients with ILD to support future studies into the development of such biomarkers. Patients with pneumonia and healthy patients will also be recruited as a control group.

DETAILED DESCRIPTION:
The proposed biospecimen repository would be derived from patients diagnosed with ILD. This is to include 500 patients in the repository, with each patient contributing one blood sample. Patients with pneumonia and healthy patients will also be recruited as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ILD or any fibrotic disease of the lung or a diagnosis of pneumonia
* Patients willing to provide written informed consent

Exclusion Criteria:

* Unwillingness/unable to give blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of ILD or any fibrotic disease of the lung. A diagnosis of pneumonia and healthy volunteers will also be included as a control group.
Sampling Method: Probability Sample
Enrollment: 635 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Future Disease Management | 1 visit
  Reliable biomarkers to help guide treatment in ILD would be a major step forward in the management of this disease.

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Carmona Porquera, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared at this time, but it may be possible that in the future outside institutions or other researchers within the Mayo Clinic may ask for specimen samples. If a specimen sample is requested, a new protocol will be submitted to the IRB or the IRB application for this study will be amended.